CLINICAL TRIAL: NCT00217165
Title: Taurine as an Anti-manic Agent: a Double-blind Placebo-controlled Study.
Brief Title: Taurine as an Anti-Manic Agent: A Double-Blind, Placebo-Controlled Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mclean Hospital (Other)
Responsible Party: Principal Investigator, Beth L. Murphy MD, PhD, Principal Investigator, Mclean Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2004P-002669
Record Dates: First submitted 2005-08-22; First posted 2005-09-22 (Estimated); Last update posted 2019-03-01 (Actual); Status verified 2019-02

CONDITIONS: Bipolar Disorder; Mania; Bipolar Depression
Keywords: bipolar; mania; depression; taurine; alternative
MeSH Terms: conditions — Bipolar Disorder; Mania; Depression | interventions — Taurine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo (Placebo Comparator): cellulose
  Interventions: Drug: taurine
- active drug (Active Comparator): taurine
  Interventions: Drug: taurine

INTERVENTIONS:
Drug: taurine — taurine 2mg BID po

SUMMARY:
The purpose of this study is to determine whether the amino acid taurine has effects on mood stability in bipolar disorder.

DETAILED DESCRIPTION:
Taurine is an amino acid that has some actions similar to mood stabilizers. Taurine is widely sold as a component of over-the-counter mood enhancing agents. However, controlled studies examining the mood effects of taurine are limited. An initial study in this laboratory looked at taurine's mood effects in individuals with bipolar disorder. This follow-up study is designed to further examine taurine's effects on manic symptoms. Subjects in the current follow-up study will add taurine or placebo to their current treatment regimen. Both depressive and manic symptoms will be tracked for three months to determine whether the addition of taurine affects mood symptoms.

ELIGIBILITY:
Inclusion Criteria:

bipolar disorder, type I bipolar disorder, type II mania hypomania mixed manic symptoms

Exclusion Criteria:

significant medical or psychiatric co-morbidity pregnancy or planning pregnancy current substance abuse or dependence

-

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2005-04; Primary Completion 2010-01 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Scores on standardized measures of manic and depressive symptoms (HAM-D, MADRS, YMRS) | 12 weeks
  MADRS and YMRS

SECONDARY OUTCOMES:
Side-effect ratings, general health ratings | 12 weeks
  SF36
Drop-outs due to medication changes | 12 weeks
  subjects leaving study before completion

CONTACTS AND LOCATIONS:
Overall Officials: Beth L Murphy, MD, PhD, Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States